CLINICAL TRIAL: NCT02087033
Title: A Randomized, Double-blinded, Cross-over Study on the Use of Ritmonutra, a Nutraceutical Product Composed of Omega 3 Fatty Acids, Astaxanthin, Vitamin E and Hawthorn in Subjects Affected by Supraventricular Ectopic Beats Without Structural Heart Disease
Brief Title: Use of Ritmonutra in Subjects Affected by Supraventricular Ectopic Beats Without Structural Heart Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is halted prematurely by sponsoring organization.
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RN-tvg-00313b
Record Dates: First submitted 2014-03-03; First posted 2014-03-14 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Arrhythmia
Keywords: supraventricular ectopic beats
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ritmonutra (Experimental): ritmonutra 2 tablets/day by mouth for 4 weeks sugar pill manufatured to simulate ritmonutra: 2 tablets/day by mouth for 4 weeks
  Interventions: Dietary Supplement: ritmonutra
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ritmonutra — 2 tablets a day by mouth for 4 weeks
  Other Names: ritmonutra rottapharm
  Arms: ritmonutra
Dietary Supplement: placebo — sugar pill manufactured to simulated ritmonutra: 2 tablets a day for 4 weeks
  Arms: placebo

SUMMARY:
it is a prospective, randomized, double-blinded, crossover study on the use of an association of omega 3 fatty acids, astaxanthin, vitamin E and hawthorn (ritmonutra) in subject affected by symptomatic supraventricular ectopic beats without structural heart disease.

The study will evaluate the reduction of the number of supraventricular ectopic beats and symptoms related.

DETAILED DESCRIPTION:
24 subjects without structural heart disease with a minimum of 300 supraventricular ectopic beats in 24 hours will be enrolled in the two participating centers and randomized to the treatment or to the placebo for 4 weeks. At the end of the first treatment period, a 24 hours Holter ECG will be performed. After 1 week of wash-out therapy, subjects will be crossed over to the other treatment for 4 weeks. Another 24 hours Holter ECG will be performed at the end of the study. During the baseline visit and during each follow up visit, symptom score and quality of life questionnaires will be completed by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 80 years
* symptomatic supraventricular ectopic beats (at least 300 in 24 hours recording)
* no structural heart disease evaluated with ecg, echocardiography, stress test and chest x-ray.
* no antiarrhythmic drug in use.

Exclusion Criteria:

* acute systemic illness
* preexcitation
* 3 or more consecutive ectopic beats
* vascular disease
* diabetes
* asthma
* soy allergy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy in reduction of supraventricular ectopic beats | 4 weeks of treatment
  the primary outcome will evaluate the reduction of the number of supraventricular ectopic beats after 4 weeks of treatment using a 24 h holter recording.

SECONDARY OUTCOMES:
Efficacy in reduction of symptoms related to supraventricular ectopic beats | 4 weeks
  the secodary outcome will evaluate the reduction of symptoms related to supraventricular ectopic beats using a symptom score and a quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: riccardo cappato, MD, Principal Investigator — Policlinico San Donato
Locations (2):
- Italy (2):
  - Policlinico San Pietro, Ponte San Pietro, Bergamo
  - Policlinico San Donato, San Donato Milanese, Milan